CLINICAL TRIAL: NCT01110876
Title: Phase I / II Adaptive Randomized Trial of Vorinostat, Erlotinib and Temozolomide in Adults With Recurrent Glioblastoma Multiforme
Brief Title: Phase I / II Vorinostat, Erlotinib and Temozolomide for Recurrent Glioblastoma Multiforme (GBM)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unanticipated Toxicities
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0651; NCI-2011-00469 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Results first posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Brain Cancer; Glioblastoma Multiforme
Keywords: Recurrent Glioblastoma Multiforme; GBM; Brain; Central Nervous Center; Malignant glioma; Glioblastoma multiforme; Gliosarcoma; Anaplastic astrocytoma; Anaplastic oligodendroglioma; Anaplastic oligoastrocytoma; Vorinostat; SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza; Erlotinib; Erlotinib Hydrochloride; OSI-774; Tarceva; Temozolomide; Temodar
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Glioma; Gliosarcoma; Astrocytoma; Oligodendroglioma | interventions — Vorinostat; Erlotinib Hydrochloride; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase I Group 1: Vorinostat + Erlotinib + Temozolomide (Experimental): Phase I 3-Drug Combination Vorinostat with Erlotinib + Temozolomide
  Starting doses Vorinostat 200 mg orally twice daily on Days 1-7 and 15-21 of every cycle; Erlotinib 200 mg orally once daily on Days 1-21; Temozolomide 125 mg/m^2 orally once daily on Days 1-7 and 15-21.
  Interventions: Drug: Vorinostat; Drug: Erlotinib; Drug: Temozolomide
- Phase I Group 2: Vorinostat + Erlotinib (Experimental): This Phase I arm to be activated only after completion of Part A of the Phase II trial of the 3-Drug combination. If part A of the Phase II trial shows lack of efficacy, trial will be terminated.
  Vorinostat orally twice daily, Days 1-14; and Erlotinib orally once daily Days 1-21 of every cycle.
  Interventions: Drug: Vorinostat; Drug: Erlotinib
- Phase II Part A 3-Drug Combination (Experimental): Vorinostat+Erlotinib+Temozolomide where drug dosing based on the MTD identified in the Phase I portion of the study.
  Vorinostat 200 mg orally twice daily on Days 1-7 and 15-21 of every cycle; Erlotinib 200 mg orally once daily on Days 1-21; Temozolomide 100 mg/m^2 orally once daily on Days 1-7 and 15-21.
  Interventions: Drug: Vorinostat; Drug: Erlotinib; Drug: Temozolomide
- Phase II Part B 2-Drug Combination (Experimental): This Phase II Part B arm to be activated only after completion of Part A of the Phase I and II Part A trial of the 3-Drug combination. If part A of the Phase II trial shows lack of efficacy, trial will be terminated.
  Vorinostat orally twice daily, Days 1-14; and Erlotinib orally once daily Days 1-21 of every cycle.
  Interventions: Drug: Vorinostat; Drug: Erlotinib

INTERVENTIONS:
Drug: Vorinostat — Phase I Starting Dose: 200 mg twice daily by mouth on Days 1-7, 15-21 of each 28 day cycle.
  Phase II Dose: MTD from Phase I.
  Other Names: SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza
Drug: Erlotinib — Phase I Starting Dose: 200 mg by mouth daily on Days 1-21 of 28 day cycle. For patients on enzyme inducing anticonvulsants (EIACs), starting dose of 400 mg.
  Phase II Dose: MTD from Phase I.
  Other Names: Erlotinib Hydrochloride; OSI-774; Tarceva
Drug: Temozolomide — 125 mg/m2 by mouth daily on days 1-7, 15-21 of each 28 day cycle.
  Other Names: Temodar
  Arms: Phase I Group 1: Vorinostat + Erlotinib + Temozolomide; Phase II Part A 3-Drug Combination

SUMMARY:
Phase I Objectives:

-To determine the maximum tolerated dose (MTD) of vorinostat + erlotinib versus vorinostat + erlotinib + temozolomide in adult patients with recurrent glioblastoma multiforme (GBM) and anaplastic gliomas.

Phase II Objectives:

Primary: To determine the efficacy of vorinostat + erlotinib versus vorinostat + erlotinib + temozolomide in patients with recurrent glioblastoma multiforme as progression free survival using a two arm adaptive randomization phase II trial design.

Secondary: To determine the radiological response, progression free survival (PFS) at 6 months, overall survival and unexpected toxicity in the two treatment arms; and to obtain exploratory data regarding histone 3 and 4 acetylation, treatment related changes in the epidermal growth factor receptor (EGFR) pathway proteins, and changes in e-cadherin and vimentin expression (mRNA /protein) levels in tumor tissue and peripheral monocytes in a subset of surgical patients.

DETAILED DESCRIPTION:
Phase I:

The Study Drugs:

Vorinostat is designed to cause chemical changes in different groups of proteins that are attached to DNA (the genetic material of cells), which may slow the growth of cancer cells or cause the cancer cells to die.

Erlotinib is designed to block the activity of a protein found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing.

Temozolomide is designed to kill cancer cells by damaging DNA (the genetic material of cells). The damaged DNA may cause tumor cell death.

Study Groups:

There are 2 phases to this study.

If you are found to be eligible to take part in the Phase I portion of this study, you will be assigned to 1 of 2 groups based on when you join this study. You will remain in the same group for the entire study. In this study, the dose level of the study drugs is different from group to group. Up to 4 dose levels of study drug combinations will be tested in Group 1, up to 2 dose levels in Group 2. Three (3) participants will be enrolled at each dose level. The first 3 participants in each group will receive the lowest dose level. Each 3 new participants will receive a higher dose than the one before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of study drugs given in combination is found.

* If you are in Group 1, you will take vorinostat, erlotinib, and temozolomide.
* If you are in Group 2, you will take vorinostat and erlotinib.

In addition, no matter which group or dose level you are assigned to, if you are on enzyme inducing anti-seizure drug, you will take a higher dose of erlotinib.

Study Drug Administration:

Each study cycle is 28 days.

If you are in Group 1:

* On Days 1-7 and 15-21 of every cycle, you will take vorinostat by mouth 2 times a day. You should take vorinostat with food. Do not open, crush, or chew the capsules.
* On Days 1-21 of every cycle, you will take erlotinib by mouth 1 time a day. You should take erlotinib in the morning 1 hour before or 2 hours after food with 1 cup (about 8 oz.) of water.
* On Days 1-7 and 15-21of every cycle, you will take the temozolomide by mouth 1 time a day. You should swallow the temozolomide capsules whole, one right after the other, without chewing them. If you vomit while taking temozolomide, you cannot take more capsules before the next scheduled dose. They should be taken on an empty stomach (at least 1 hour before and 2 hours after eating) with 1 cup (about 8 ounces) of water.

If you are in Group 2:

* On Days 1-14 of every cycle, you will take vorinostat by mouth 2 times a day. You should take vorinostat with food. Do not open, crush, or chew the capsules.
* On Days 1-21 of every cycle, you will take erlotinib by mouth 1 time a day. You should take erlotinib in the morning 1 hour before or 2 hours after food with 1 cup (about 8 oz.) of water.

Study Visits:

Every 4 weeks for the first 8 weeks, then every 8 weeks after that:

* Your complete medical history will be recorded.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a neurological exam.
* Your performance status will be recorded.

Every week for the first 4 weeks, then every 2 weeks after that, blood (about 3 teaspoons) will be drawn for routine tests and to check your blood's ability to clot normally.

Every 4 weeks, if you are on anti-seizure drugs, blood (about 1 teaspoon) will be drawn to measure the amount of anti-seizure drugs in your blood.

Every 8 weeks, you will have an MRI scan to check the status of the disease.

Length of Study:

You will be on study for up to 1 year. You may continue to receive the study drugs beyond 1 year and remain on study if your doctor decides that it is in your best interest. You will be taken off study early if the disease gets worse or you experience intolerable side effects.

Long-Term Follow-Up Visit:

If you go off study after 12 cycles, blood (about 3 teaspoons) will be drawn for routine tests and to check your blood's ability to clot normally every 2 weeks during the 30 days after your last dose of study drugs.

If you go off the study for reasons other than the worsening of the disease, you will have an MRI every 2 months unless the disease gets worse.

If you have an MRI that shows worsening of the disease, every 2-3 months from then on, you may be called and asked how you are feeling and about any new cancer treatment that you may have received. This phone call should take about 5-10 minutes.

This is an investigational study. Erlotinib is FDA approved drug for treatment of some types of non-small cell lung cancer, temozolomide for some types of brain cancer, and vorinostat for some types of lymphoma. All are commercially available. The use of these drugs in this combination is investigational.

Up to 182 participants will take part in this study. Up to 72 patients will be enroll in the Phase 1 portion of this study. All will be enrolled at MD Anderson.

Phase II:

The Study Drugs:

Vorinostat is designed to cause chemical changes in different groups of proteins that are attached to DNA (the genetic material of cells), which may slow the growth of cancer cells or cause the cancer cells to die.

Erlotinib is designed to block the activity of a protein found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing.

Temozolomide is designed to kill cancer cells by damaging DNA (the genetic material of cells). The damaged DNA may cause tumor cell death.

Study Groups:

There are 2 phases to this study.

If you are found to be eligible to take part in the Phase 2 portion of this study, you will be randomly assigned (as in the roll of the dice) to 1 of 2 groups.

* If you are in Group 1, you will take vorinostat and erlotinib.
* If you are in Group 2, you will take vorinostat, erlotinib, and temozolomide.

Subset Group:

If your doctor has recommended that you have surgery to remove a tumor that has come back, you will be eligible for this subset group. You would have the surgery before being assigned to a main study group. This subset group of the study is done to learn the effects of vorinostat on tumor tissue and blood cells.

Before surgery, you will be randomly assigned to 1 of 3 groups.

* If you are in Group A, you will receive vorinostat alone.
* If you are in Group B, you will receive erlotinib alone.
* If you are in Group C, you will receive both vorinostat and erlotinib.

You will take the study drug(s) for 3 days in a row before your surgery.

About 2 weeks after the surgery, you will be randomly assigned to 1 of 2 main study groups described above (Group 1 or 2).

In addition, no matter which group you are assigned to, if you are on enzyme inducing anti-seizure drug, you will take the higher dose of erlotinib.

Study Drug Administration:

Every cycle is 28 days.

If you are in Group 1:

* On Days 1-14 of every cycle, you will take vorinostat by mouth 2 times a day. You should take vorinostat with food. Do not open, crush, or chew the capsules.
* On Days 1-21 of every cycle, you will take erlotinib by mouth 1 time a day. You should take erlotinib in the morning 1 hour before or 2 hours after food with 1 cup (about 8 oz.) of water.

If you are in Group 2:

* On Days 1-7 and 15-21 of every cycle, you will take vorinostat by mouth 2 times a day .You should take vorinostat with food. Do not open, crush, or chew the capsules.
* On Days 1-21 of every cycle, you will take erlotinib by mouth 1 time a day . You should take erlotinib in the morning 1 hour before or 2 hours after food with 1 cup (about 8 oz.) of water.
* On Days 1-7 and 15-21 of every cycle, you will take the temozolomide by mouth 1 time a day. You should swallow the temozolomide capsules whole, one right after the other, without chewing them. If you vomit while taking temozolomide, you cannot take more capsules before the next scheduled dose. They should be taken on an empty stomach (at least 1 hour before and 2 hours after eating) with 1 cup (about 8 ounces) of water.

Subset group:

For 3 days in row before surgery:

* If you are in Group A, you will take vorinostat by mouth 2 times a day.
* If you are in Group B, you will take erlotinib by mouth 1 time a day.
* If you are in Group C, you will take vorinostat by mouth 2 time a day and erlotinib by mouth 1 time a day.

After you have recovered from the effects of surgery (about 2 weeks), you will follow the study group schedule (Group 1 or 2) described above.

Study Visits:

Every 4 weeks for the first 8 weeks, then every 8 weeks after that:

* Your complete medical history will be recorded.
* You will be asked about any drugs you may be taking and if you have had any side effects.
* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a neurological exam.
* Your performance status will be recorded.

Every week for the first 4 weeks, then every 2 weeks after that, blood (about 3 teaspoons) will be drawn for routine tests and to check your blood's ability to clot normally.

Every 4 weeks, if you are on anti-seizure medications, blood (about 1 teaspoon) will be drawn to measure the amount of anti-seizure medications in your blood.

Every 8 weeks, you will have an MRI scan to check the status of the disease.

Subset Group:

In addition to the above tests, blood (about 1 teaspoon each time) will be drawn 1 time before and 3 times after the first dose of vorinostat, and during surgery. This blood will be used to study the drug levels, the effects of the drug in normal blood cells, and to match these findings with that in the tumor.

After the surgery, part of the leftover tumor tissue from the surgery will be used to measure the drug levels and the effects of vorinostat on the tumor and be used for biomarker tests.

Length of Study:

You will be on study for up to 1 year. You may continue to receive treatment beyond 1 year and remain on study if your doctor decides that it is in your best interest. You will be taken off study early if the disease gets worse or you have intolerable side effects.

Long-Term Follow-Up Visit:

If you go off study after 12 cycles, blood (about 3 teaspoons) will be drawn for routine tests and to check your blood's ability to clot normally every 2 weeks during the 30 days after your last dose of study drugs.

If you go off the study for reasons other than the worsening of the disease, you will have an MRI every 2 months unless the disease gets worse.

If you have an MRI that shows worsening of the disease, every 2-3 months from then on, you may be called and asked how you are feeling and about any new cancer treatment that you may have received. This phone call will take about 5-10 minutes.

This is an investigational study. Erlotinib is FDA approved drug for treatment of some types of non-small cell lung cancer, temozolomide for some types of brain cancer, and vorinostat for some types of lymphoma. All are commercially available. The use of these drugs in this combination is investigational.

Up to 182 participants will take part in this study. Up to 110 patients will be enrolled in the Phase 2 portion of this study. Up to 15 participants will take part in the subset portion of the study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven glioblastoma multiforme, gliosarcoma or anaplastic glioma will be eligible for the Phase I component. Anaplastic gliomas include anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic oligoastrocytoma (AOA), or malignant glioma not otherwise specified (NOS). Patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a malignant glioma is made. Only patients with histologically proven supratentorial glioblastoma multiforme or gliosarcoma will be eligible for the Phase II component.
2. Patients must have shown unequivocal evidence for tumor recurrence or progression by MRI scan and should have failed radiation therapy. Patients should have completed radiation therapy at least 3 months prior to entry into the study. The scan done prior to study entry documenting progression will be reviewed by the treating physician to document changes in tumor dimension to confirm recurrence.
3. (2. continued) Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have reasonable confirmation of true progressive disease rather than radiation necrosis as determined by the treating physician and neuro-radiologist; for example, through MRI, magnetic resonance (MR) spectroscopy, or PET scan of the brain.
4. For the Phase I component, any number of prior relapses is allowed, provided the patient fulfills all other eligibility criteria particularly that of the functional status. For the phase II component, patients may have had up to 2 prior relapses
5. All patients must sign an informed consent indicating their awareness of the investigational nature of this study in keeping with the policies of this hospital.
6. The baseline on-study MRI should be performed within 14 days (+/- 3 days) prior to registration and on a steroid dosage that has been stable or decreasing for at least 5 days. If the steroid dose is increased between the date of imaging and the initiation of therapy (or at that time), a new baseline MRI is required. The same type of scan, i.e., MRI, must be used throughout the period of protocol treatment for tumor measurement.
7. Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply: a) They have recovered from the effects of surgery. b) Evaluable or measurable disease following resection of recurrent tumor is not mandated for eligibility into the study. c) To best assess the extent of residual measurable disease post-operatively, a MRI should be done no later than 96 hours in the immediate post-operative period or 4-6 weeks post-operatively.
8. Patients must be 18 years old or older.
9. Patients must have a Karnofsky performance status (KPS) equal or greater than 60
10. Patients must have recovered from the toxic effects of prior therapy to grade 1 non hematological or </= grade 2 hematological toxicity (except deep vein thrombosis): 4 weeks from prior cytotoxic therapy or bevacizumab and/or at least two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, cis-retinoic acid, etc. (radiosensitizer does not count).
11. (10. continued) Patients who receive anticancer agents for non-therapeutic purposes unrelated to this study (such as presurgically for obtaining pharmacology data for the agent) will be eligible to enter the study provided they have recovered from the toxic effects of the agent if any. Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.
12. Patients must have adequate bone marrow function (ANC>/= 1,500/mm^3 and platelet count of >/= 100,000/mm^3), adequate liver function (SGPT </= 3 times normal and alkaline phosphatase </= 2 times normal, bilirubin </= 1.5 mg/dl), adequate renal function (BUN and creatinine </= 1.5 times institutional normal) prior to registration.
13. Women of childbearing potential on treatment must not be pregnant, must not be breast-feeding and must practice adequate contraception. Male patients on treatment with vorinostat must agree to use an adequate method of contraception for the duration of the study, and for 30 days after the last dose of study medication.

Exclusion Criteria:

1. Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix or bladder), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
2. Patients must not have: a) active infection b) disease that will obscure toxicity or dangerously alter drug metabolism, especially liver disease including cirrhosis or hepatic dysfunction c) serious intercurrent medical illness
3. Patients who are currently on active treatment for AIDS or hepatitis will be excluded due to the potential for adverse interaction with ongoing treatment agents and for unknown toxicity.
4. Patients receiving valproic acid (VPA), an anticonvulsant drug with histone deacetylase (HDAC) inhibitor properties, will be excluded, unless they are switched to an alternative agent prior to treatment initiation. A 5 day wash out period is required.
5. Prior treatment with EGFR inhibitors or temozolomide on a standard day 1-5 dosing and low dose daily dosing as part of chemoradiation therapy is allowed because the trial is based on the hypothesis that the combination of agents used will be synergistic in their effects, and that HDAC inhibition will potentially overcome resistance to EGFR inhibitors and temozolomide. However, prior treatment with dose dense regimens of temozolomide (7 days on/ 7 days off, 21 days/28 days or continuous low dose daily dosing not with chemoradiation) and HDAC inhibitors other than valproic acid (such as depsipeptide, LBH-589 or vorinostat) are not permitted.
6. Patients with a known allergy to any component of vorinostat, or a known allergy to Temozolomide or erlotinib will be excluded.
7. Patient must be able to tolerate the procedures required in this study including periodic blood sampling, study related assessments, and management at the treating institution for the duration of the study. Inability to comply with protocol or study procedures (for example, an inability to swallow tablets) will be an exclusion criteria.
8. This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender.
9. No exclusion to this study will be based on race. The malignant glioma patient population treated at MD Anderson Cancer Center (MDACC) over the past year is as follows: American Indian or Alaskan Native - 0; Asian or Pacific Islander - <2%; Black, not of Hispanic Origin - 3%; Hispanic - 6%; White, not of Hispanic Origin - 88%; Other or Unknown - 2%; Total-100%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John DeGroot, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 21, 2011 to March 18, 2013. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 14 participants registered in Phase I, two participants did not begin study due to financial reasons and were excluded. One of the six participants in Phase II one was not eligible and is also excluded. The study did not progress to the next stage of Phase II with adaptive randomized arms.
Groups:
- Phase I: Vorinostat + Erlotinib + Temozolomide: Phase I 3-Drug Combination Vorinostat with Erlotinib + Temozolomide
  Starting doses Vorinostat 200 mg orally twice daily on Days 1-7 and 15-21 of every cycle; Erlotinib 200 mg orally once daily on Days 1-21; Temozolomide 125 mg/m^2 orally once daily on Days 1-7 and 15-21.
Period: Overall Study
Arm/Group | Phase I: Vorinostat + Erlotinib + Temozolomide | Phase II Part A 3-Drug Combination
Started | 13 (One received 400 mg Erlotinib dose as result of enzyme inducing anticonvulsants (EIACs)) | 5
Completed | 13 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I Group 1: Vorinostat + Erlotinib + Temozolomide: Phase I 3-Drug Combination Vorinostat with Erlotinib + Temozolomide
  Starting doses Vorinostat 200 mg orally twice daily on Days 1-7 and 15-21 of every cycle; Erlotinib 200 mg orally once daily on Days 1-21; Temozolomide 125 mg/m2 orally once daily on Days 1-7 and 15-21.
- Phase II Part A 3-Drug Combination: Vorinostat+Erlotinib+Temozolomide where drug dosing based on the MTD identified in the Phase I portion of the study.
  Vorinostat 200 mg orally twice daily on Days 1-7 and 15-21 of every cycle; Erlotinib 200 mg orally once daily on Days 1-21; Temozolomide 100 mg/m2 orally once daily on Days 1-7 and 15-21.
- Total: Total of all reporting groups
Arm/Group | Phase I Group 1: Vorinostat + Erlotinib + Temozolomide | Phase II Part A 3-Drug Combination | Total
Number analyzed (Participants) | 13 | 5 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 4 | 16
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Full Range); unit: years] | 48 [28 to 73] | 53 [42 to 67] | 51 [28 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 13 | 5 | 18
Enzyme Inducing Anti-Convulsants (EIACs) [Count of Participants; unit: Participants]
  EIACs | 1 | 0 | 1
  NEIACs | 12 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Vorinostat in Combination With Escalating Doses of Erlotinib and Temozolomide
Description: Phase I assessment MTD Vorinostat in combination with escalating doses of Erlotinib and Temozolomide using conventional phase I design where 3 enrolled into first dose level, monitored for 3 weeks and if no dose-limiting toxicity (DLT) seen, 3 more enrolled at next dosage level. If 2/6 participants experience DLT, the previous (lower) dosage level declared MTD of vorinostat in combination with Erlotinib and Temozolomide.
  A maximum of 4 dosage levels utilized with deescalation by 2 dose levels if DLT is seen at the starting dose level. If no DLT noted after dose escalation to Level 4, these doses utilized as MTD for phase II.
Time Frame: Evaluated with each 28 day (+2 days) cycle, up to 24 weeks
Population: One participant started later than 12 assigned to original MTD dose levels, and was excluded from this analysis.
Measure: Number; unit: mg
Arm/Group | Phase I Group 1: Vorinostat + Erlotinib + Temozolomide
Number analyzed (Participants) | 12
mg
  Vorinostat (mg) twice/day | 200
  Erlotinib (mg) | 200

2. Secondary Outcome: Progression Free Survival (PFS)
Description: This is an adaptive randomized phase II trial to Vorinostat + Erlotinib to Vorinostat + Erlotinib + Temozolomide in patients with recurrent GBM. The primary outcome is progression free survival (PFS). Patients will be randomized between the two arms using a Bayesian adaptive algorithm. Participants randomized equally between the two arms at the start of the trial (for the first 20 patients). Thereafter, as the trial progresses and data accrue, the randomization will become unbalanced in favor of the treatment that, on average, has better results in terms of failure time. Therefore, each successive patient is more likely to receive the treatment with better results, on average.
Time Frame: 6 months
Population: No data collected. The study did not progress to the next stage of Phase II with adaptive randomized arms.
Arm/Group | Phase I Group 1: Vorinostat + Erlotinib + Temozolomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection events that occurred after participants received study drug through a treatment cycle of 28 days (+3 days) and within 30 days of last treatment dose.
Description: Due to effect enzyme inducing anticonvulsants (EIACs) on erlotinib, 2 different Phase I dosing schedules (participants on EIACs or those on non-enzyme inducing antiepileptics (NEIACs) were used. AEs reported separately. Participants experiencing different adverse events with different grade are counted only once at highest grade experienced.
Groups:
- Phase I Dose 0: Vorinostat 200 mg + Temozolomide 125 mg/m^2: Phase I 3-Drug Combination Vorinostat with Erlotinib + Temozolomide
  Vorinostat 200 mg orally twice daily on Days 1-7 and 15-21 of every cycle; Erlotinib 200 mg orally once daily on Days 1-21; Temozolomide 125 mg/m^2 orally once daily on Days 1-7 and 15-21.
- Phase I Dose -1: Vorinostat 200 mg + Temozolomide 100 mg/m^2: Phase I 3-Drug Combination Vorinostat with Erlotinib + Temozolomide
  Vorinostat 200 mg orally twice daily on Days 1-7 and 15-21 of every cycle; Erlotinib 200 mg twice daily on Days 1-21; Temozolomide 100 mg/m^2 orally once daily on Days 1-7 and 15-21.
- Phase I EIACs: Vorinostat 400 mg + Temozolomide 125 mg/m^2: Phase I 3-Drug Combination Vorinostat with Erlotinib + Temozolomide for participant on enzyme inducing anticonvulsants (EIACs):
  Vorinostat 400 mg orally twice daily on Days 1-7 and 15-21 of every cycle; Erlotinib 100 mg orally once daily on Days 1-21; Temozolomide 125 mg/m^2 orally once daily on Days 1-7 and 15-21.
- Phase II 3-Drug Combination: Vorinostat+Erlotinib+Temozolomide where drug dosing based on the MTD identified in the Phase I portion of the study.
  Vorinostat 200 mg orally twice daily on Days 1-7 and 15-21 of every cycle; Erlotinib 200 mg orally once daily on Days 1-21; Temozolomide 100 mg/m^2 orally once daily on Days 1-7 and 15-21.
Arm/Group | Phase I Dose 0: Vorinostat 200 mg + Temozolomide 125 mg/m^2 | Phase I Dose -1: Vorinostat 200 mg + Temozolomide 100 mg/m^2 | Phase I EIACs: Vorinostat 400 mg + Temozolomide 125 mg/m^2 | Phase II 3-Drug Combination
Serious Adverse Events (participants affected / at risk) | 3/6 | 4/6 | 0/1 | 1/5
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 1/1 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose 0: Vorinostat 200 mg + Temozolomide 125 mg/m^2 (N=6) | Phase I Dose -1: Vorinostat 200 mg + Temozolomide 100 mg/m^2 (N=6) | Phase I EIACs: Vorinostat 400 mg + Temozolomide 125 mg/m^2 (N=1) | Phase II 3-Drug Combination (N=5)
Death (General disorders) | 1 | 0 | 0 | 0
BILIRUBIN (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Central Nervous System (CNS) ISCHEMIA (Nervous system disorders) | 0 | 2 | 0 | 0
DEHYDRATION (Gastrointestinal disorders) | 0 | 2 | 0 | 0
DIARRHEA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
FATIGUE (General disorders) | 0 | 1 | 0 | 0
HYPONATREMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
INFECTION CLINICAL (Infections and infestations) | 0 | 1 | 0 | 0
MENTAL STATUS (Nervous system disorders) | 1 | 0 | 0 | 0
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0
PLATELETS, DECREASE (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
SEIZURE (Nervous system disorders) | 1 | 2 | 0 | 0
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 0 | 1 | 0 | 0
Neurological Disorder (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose 0: Vorinostat 200 mg + Temozolomide 125 mg/m^2 (N=6) | Phase I Dose -1: Vorinostat 200 mg + Temozolomide 100 mg/m^2 (N=6) | Phase I EIACs: Vorinostat 400 mg + Temozolomide 125 mg/m^2 (N=1) | Phase II 3-Drug Combination (N=5)
ACNE (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0
ALKALINE PHOSPHATASE (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
ALLERGIC RHINITIS (Immune system disorders) | 1 | 0 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
ALT SGPT (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0
ANOREXIA (Gastrointestinal disorders) | 3 | 3 | 1 | 0
AST SGOT (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0
BICARBONATE SERUM-LOW (Metabolism and nutrition disorders) | 3 | 4 | 0 | 0
BILIRUBIN (Blood and lymphatic system disorders) | 5 | 4 | 0 | 3
BLURRED VISION (Eye disorders) | 0 | 0 | 1 | 0
CNS ISCHEMIA (Nervous system disorders) | 0 | 2 | 0 | 0
COGNITIVE DISTURBANCE (Psychiatric disorders) | 0 | 0 | 1 | 0
CONFUSION (Psychiatric disorders) | 2 | 4 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 2 | 1 | 1 | 2
CREATININE (Metabolism and nutrition disorders) | 5 | 3 | 0 | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
DEHYDRATION (Gastrointestinal disorders) | 1 | 2 | 0 | 0
DIARRHEA (Gastrointestinal disorders) | 6 | 6 | 1 | 3
DIZZINESS (Nervous system disorders) | 0 | 2 | 0 | 1
DRY MOUTH (Gastrointestinal disorders) | 1 | 2 | 1 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 2 | 0 | 0
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
FATIGUE (General disorders) | 4 | 4 | 1 | 5
FEVER WITHOUT NEUTROPENIA (General disorders) | 1 | 1 | 0 | 0
GAIT/WALKING (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0 | 0
HEARING (W/O MONITORING) (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
HEARTBURN (Gastrointestinal disorders) | 0 | 1 | 1 | 0
HEMOGLOBIN (Blood and lymphatic system disorders) | 5 | 4 | 1 | 3
HEMORRHAGE GU (KIDNEY) (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
HEMORRHAGE PULMONARY (NOSE) (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
HEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
HICCOUGHS (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 | 4 | 0 | 3
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPERTENSION (Cardiac disorders) | 0 | 1 | 0 | 0
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 2 | 3 | 0 | 2
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 | 3 | 0 | 2
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
HYPOKALEMIA (Metabolism and nutrition disorders) | 4 | 2 | 0 | 3
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
HYPONATREMIA (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0
INCONTINENCE URINARY (Renal and urinary disorders) | 0 | 1 | 0 | 1
INFECTION CLINICAL + GRADE 3-4 ANC (URINARY TRACT NOS) (Infections and infestations) | 1 | 1 | 0 | 0
INFECTION UNKNOWN ANC (URINARY TRACT NOS) (Infections and infestations) | 2 | 0 | 0 | 0
INFECTION W NORMAL ANC (UPPER AIRWAY NOS) (Infections and infestations) | 1 | 0 | 1 | 1
INFECTION W NORMAL ANC (URINARY TRACT NOS) (Infections and infestations) | 3 | 2 | 0 | 0
INFECTION W NORMAL ANC(BLOOD SEPSIS) (Infections and infestations) | 1 | 0 | 0 | 0
INSOMNIA (General disorders) | 1 | 0 | 1 | 0
LEUKOCYTES (Blood and lymphatic system disorders) | 4 | 3 | 1 | 0
LIPASE INCREASED (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 5 | 4 | 1 | 4
MEMORY IMPAIRMENT (Psychiatric disorders) | 0 | 3 | 1 | 0
MENTAL STATUS (Psychiatric disorders) | 1 | 0 | 0 | 0
METABOLIC/LABORATORY (OTHER) (Metabolism and nutrition disorders) | 5 | 5 | 0 | 4
MOOD ALTERATION (DEPRESSION) (Psychiatric disorders) | 0 | 1 | 1 | 0
MUCOSITIS (SYMPTOMATIC) ORAL CAVITY (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1 | 0
MUSCLE WEAKNESS (LEFT-SIDED) (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
MUSCLE WEAKNESS (WHOLE BODY/GENERALIZED) (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 3
MUSCULOSKELETAL (OTHER) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
NASAL/PARANASAL REACTIONS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 6 | 4 | 1 | 1
NEUROLOGY (OTHER) (Psychiatric disorders) | 1 | 1 | 0 | 2
NEUTROPHILS (ANC/AGC) (Blood and lymphatic system disorders) | 3 | 3 | 0 | 0
OCULAR/VISUAL (OTHER) (Eye disorders) | 1 | 0 | 0 | 0
PAIN (ABDOMEN NOS) (General disorders) | 0 | 2 | 1 | 0
PAIN (BACK) (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
PAIN (CHEST/THORAX) (General disorders) | 1 | 1 | 0 | 0
PAIN (EXTREMITY-LIMB) (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
PAIN (HEAD/HEADACHE) (Nervous system disorders) | 3 | 3 | 1 | 1
PAIN (MUSCLE) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
PAIN (ORAL CAVITY) (Gastrointestinal disorders) | 0 | 1 | 0 | 1
PAIN (OTHER) (General disorders) | 1 | 0 | 0 | 0
PAIN (THROAT/PHARYNX/LARYNX) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PALPITATIONS (Cardiac disorders) | 0 | 1 | 1 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
PLATELETS (Blood and lymphatic system disorders) | 6 | 4 | 0 | 3
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1
PSYCHOSIS (Psychiatric disorders) | 0 | 1 | 0 | 0
PYRAMIDAL TRACT DYSFUNCTION (Nervous system disorders) | 0 | 0 | 1 | 0
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 2
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 0 | 0
RIGORS/CHILLS (General disorders) | 0 | 1 | 0 | 0
SEIZURE (General disorders) | 3 | 2 | 0 | 0
SOMNOLENCE (Psychiatric disorders) | 1 | 1 | 0 | 0
SPEECH IMPAIRMENT (Psychiatric disorders) | 2 | 4 | 1 | 0
SYNCOPE (FAINTING) (Nervous system disorders) | 1 | 0 | 0 | 1
TASTE ALTERATION (Gastrointestinal disorders) | 0 | 2 | 0 | 0
THROMBOSIS/THROMBUS/EMBOLISM (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
TREMOR (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
URINARY FREQUENCY (Renal and urinary disorders) | 0 | 1 | 0 | 0
URINE COLOR CHANGE (Renal and urinary disorders) | 1 | 0 | 0 | 0
VOICE CHANGES (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 4 | 2 | 0 | 0
WEIGHT LOSS (General disorders) | 1 | 3 | 0 | 1
BRUISING (NO THROMBOPENIA) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
CUSHINGOID (Endocrine disorders) | 0 | 0 | 0 | 1
DIPLOPIA (Eye disorders) | 0 | 0 | 0 | 1
EDEMA: LIMB (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
HYPOTENSION (Cardiac disorders) | 0 | 0 | 0 | 1
INFECTION UNKNOWN ANC (UPPER AIRWAY NOS) (Infections and infestations) | 0 | 0 | 0 | 1
INFECTION W NORMAL ANC (CONJUNCTIVA) (Infections and infestations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes